CLINICAL TRIAL: NCT01863212
Title: Investigating the Role of the FTO Gene in Reward System Activation During Visual Presentation of Food Images With fMRI Technique
Brief Title: The Role of the FTO Gene in Reward System Activation in Obese and Healthy Subjects
Acronym: FTO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: LSF008786
Record Dates: First submitted 2013-05-21; First posted 2013-05-27 (Estimated); Last update posted 2013-05-27 (Estimated); Status verified 2013-05

CONDITIONS: Obesity; Eating Behavior
MeSH Terms: conditions — Obesity; Feeding Behavior | interventions — Blood Specimen Collection; Stroop Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Risk allele carriers (Experimental): Individuals homozygous for the risk allele (A/A) The interventions administrated to this group: 'Blood sampling for genetic analyse', 'Stroop test', 'fMRI'
  Interventions: Procedure: Blood sampling for genetic analyse; Behavioral: Stroop test; Other: fMRI
- Non risk allele carriers (Experimental): Individuals homozygous for the non-risk allele (T/T) The interventions administrated to this group: 'Blood sampling for genetic analyse', 'Stroop test', 'fMRI'
  Interventions: Procedure: Blood sampling for genetic analyse; Behavioral: Stroop test; Other: fMRI

INTERVENTIONS:
Procedure: Blood sampling for genetic analyse — Blood sampling are performed at the initiation visit in order to screen for allele variants
Behavioral: Stroop test — Selective attention test where subjects, in one minute, names the ink color of several words without naming the word itself.
Other: fMRI — Functional Magnetic Resonance Imaging, performed to view brain activity

SUMMARY:
In order to investigate if individuals, carrying genetic variants predisposing to obesity, respond differently to visual presented food images than non-carriers the investigators aim to screen 500 people for a common risk variant in the FTO gene. From those 500 screened 40 subjects, 20 homozygous for the risk allele and 20 homozygous for a non risk allele will be selected for the second step in the study. This part involves the fMRI technique to visualize the brain response, focus on reward system activation, when food images are visually presented in the scanner. Factors regarding eating behavior, sleep, physical exercise and relation to food are investigated in the first part of the study as well as clinical parameters such as BMI.

ELIGIBILITY:
Inclusion Criteria:

* No medications (except contraceptives including estrogen)
* No metabolic disorders/diseases
* Right handed
* Color vision
* Normal sleep-wake rhythm (eg. shift workers can not participate)

Exclusion Criteria:

* Specific preferences of food, for example vegetarians
* Grandparents originating from country outside the Nordic area
* Metallic implants

Ages: 18 Years to 37 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 500 (Estimated)
Dates: Start 2010-09; Primary Completion 2014-09 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Genotyping for variants in the FTO gene associated with overweight and obesity | Blood sampling for genetic analyse is performed at the initiation visit

CONTACTS AND LOCATIONS:
Overall Officials: Christian Benedict, PhD, Principal Investigator — dep. Neuroscience, Uppsala University
Locations (2):
- Sweden (2):
  - Uppsala University, Uppsala, Uppsala County
  - dep. Neuroscience, Uppsala University, Uppsala, Uppsala County

REFERENCES:
- [Derived] Andreoli MF, De Francesco PN, Titova OE, Perello M, Schioth HB. Plasma LEAP2 concentration is associated with attention and cognitive responses to low-calorie food cues in men depending on body weight status. Physiol Behav. 2025 Nov 1;301:115049. doi: 10.1016/j.physbeh.2025.115049. Epub 2025 Aug 7. PMID 40759193
- [Derived] Wiemerslage L, Islam R, van der Kamp C, Cao H, Olivo G, Ence-Eriksson F, Castillo S, Larsen AL, Bandstein M, Dahlberg LS, Perland E, Gustavsson V, Nilsson J, Vogel H, Schurmann A, Larsson EM, Rask-Andersen M, Benedict C, Schioth HB. A DNA methylation site within the KLF13 gene is associated with orexigenic processes based on neural responses and ghrelin levels. Int J Obes (Lond). 2017 Jun;41(6):990-994. doi: 10.1038/ijo.2017.43. Epub 2017 Feb 14. PMID 28194012